CLINICAL TRIAL: NCT05322109
Title: Diagnostic Accuracy of Cardiac Magnetic Resonance Tomography (CMR) for Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Cardiac Magnetic Resonance Tomography for Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: German Heart Institute (Other)
Responsible Party: Principal Investigator, Sebastian Kelle, Principal Investigator, German Heart Institute
Other Study IDs: EA2/017/22
Record Dates: First submitted 2022-03-03; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure, Diastolic
Keywords: cardiac magnetic resonance; magnetic resonance imaging; lvedp
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMR — Clinically indicated cardiac magnetic resonance tomography executed according to international guideline recommendations.
  Other Names: Cardiac magnetic resonance tomography

SUMMARY:
The diagnosis of heart failure with preserved ejection fraction has so far been made primarily according to criteria determined by echocardiography, or invasively by measuring the left ventricular filling pressures. Increasingly, CMR is also evaluated with regard to the diagnosis of cardiac insufficiency with preserved pump function.However, it is still unclear which parameters can be used meaningfully for diagnostics.To answer this question, the investigators want to retrospectively evaluate data collected from patients with a clinical indication for CMR and coronary angiography.

DETAILED DESCRIPTION:
Heart failure with preserved pump function is a common disease that is associated with a high level of suffering for the patient. The diagnosis has so far been made primarily according to criteria determined by echocardiography, or invasively by measuring the left ventricular filling pressures.

With its high spatial resolution and the possibility of tissue-specific diagnostics, cardiac MRI (CMR) offers outstanding possibilities in cardiac imaging without exposing the patient to ionizing radiation. Increasingly, CMR is also evaluated with regard to the diagnosis of cardiac insufficiency with preserved pump function. However, it is still unclear which parameters can be used meaningfully for diagnostics. There is evidence for a correlation with invasively increased LVEDP, although the number of patients examined in the previous studies was still small. In addition, possible influences from medication and clinical parameters were not examined.

To answer this question, the investigators want to retrospectively evaluate data collected from patients with a clinical indication. The significance of the study is that in the future CMR could supplement echocardiography in the diagnosis of HFpEF and further reduce the need for invasive diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CMR and left heart catheterization including LVEDP measurement within the same month

Exclusion Criteria:

* Severe Valve Dysfunction or Pericardial/Pleural Disease
* Contraindictaion for CR or Cath

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: atients with CMR and left heart catheterization including LVEDP measurement within the same month
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Extracellular myocardial volume (%) | One montth
  Estimated percentage of extracellular volume of the myocardium
Left atrial volume (ml) | One month
  Volume of the left atrium in mililiters

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request anonymized IPD may be sharedn at the discretion of the PI.